CLINICAL TRIAL: NCT04871230
Title: Dried Blood Spot Test to Assess TB in Pregnancy in Remote and Resource Limited Areas
Brief Title: Dried Blood Spot Test to Assess TB in Pregnancy
Acronym: DROPTB2
Status: Completed | Type: Observational
Sponsor: Institut Pasteur de Madagascar (Other)
Collaborators: National Tuberculosis Program, Madagascar (Unknown); Analakely Hospital University Care and Public Health, Madagascar (Unknown); Virginia-Maryland College Veterinary Medecine, Blacksburg (Unknown); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01; TTS-2008-25933 (Other Grant/Funding Number: Grand Challenges Canada)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Tuberculosis
Keywords: Pregnant women; Tuberculosis; Diagnostic; Genes signature; Dried Blood Spot
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The novel test is based on measurements of relative amounts of mRNA expression associated with 3 target genes identified through a genome-wide multicohort analysis using genetic sequencing data from confirmed pulmonary TB patients. The 3-gene mRNA-based q-PCR test (3G q-PCR) is able to detect infection in 93% of patients, can differentiate between active pulmonary disease and latent infection with good sensitivity (i.e. 88%)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women suspected TB: This group enrolled as cases
  Interventions: Diagnostic Test: 3G DBS; Diagnostic Test: Sputum Test; Diagnostic Test: 3G Veinous Blood
- Pregnant women without signs suspected TB: This group enrolled as controls
  Interventions: Diagnostic Test: 3G DBS; Diagnostic Test: 3G Veinous Blood

INTERVENTIONS:
Diagnostic Test: 3G DBS — Collection of capillary blood samples for the 3G q-PCR test
  Other Names: 3G qPCR test with Dried Blot Spot Samples
Diagnostic Test: Sputum Test — Collection of sputum for test culture, microscopy, GeneXpert
  Other Names: Culture sputum; GeneXpert Sputum; Microscopy Sputum
  Groups: Pregnant women suspected TB
Diagnostic Test: 3G Veinous Blood — Collection liquid veinous blood for the 3G q-PCR test

SUMMARY:
Despite being a key contributor to maternal mortality in high-burden regions, TB in pregnancy is a hugely neglected area of global public health. During pregnancy, the symptoms of TB are often overlooked and undiagnosed because they are vague, non-specific, and can be very similar to common complaints during pregnancy. Women with TB in pregnancy are at an increased risk of anemia and perinatal death.

The DROP-TB project aims to expand the tuberculosis (TB) detection testing in pregnancy by creating a system where blood samples are collected from women at their local healthcare clinics instead of/or at national-level TB diagnostic centres where visits can require substantial travel and cost. Blood samples collected in specific RNA stabilizing tubes and on specific storing paper filters are collected from pregnant women with presumptive TB and transported to a central TB testing facility and analyzed by real-time polymerase chain reaction (qPCR).

The DROP-TB method measures the mRNA expressions known to be markers of TB infection and disease. Based on veinous blood sampling, those signatures have showed high sensitivity (93%) and specificity (97%), can differentiate between active and latent infection, and performs well in the presence of other infections such as HIV. The DROP-TB program was specifically designed to increase the coverage of TB testing in pregnancy to improve health outcomes for women and their unborn children.

The evidence generated from this program will demonstrate the feasibility of this program in providing TB diagnosis to women in rural and remote regions of LMIC with the example of Madagascar. Evidence will be presented to policy makers as a case to support the national scale up of the program in LMICs.

DETAILED DESCRIPTION:
With this Grand Challenges Canada Transition to scale DROP-TB program, the Institut Pasteur de Madagascar will:

1. Conduct a validation trial of the DROP-TB screening program in rural Madagascar, enrolling 3,500 women with presumptive TB, of which ~1,229 will be pregnant women
2. Support the development of laboratory capacity to collect veinous, DBS and other samples for qPCR at the 101 TB testing centres participating in the trial and implement standard operating procedures for DROP-TB testing
3. Assess the implementation and cost of the shipping program to bring different type of blood samples from community-based centres to national health centres for testing.

This is a cross -sectional study conducted on pregnant women suspected of having pulmonary TB (n = 1300), pregnant women without apparent pathology (controlled pregnant women), TB indemnity and without notion of tuberculous contact ( n = 50) and non -pregnant women were also free of TB and without a notion of tuberculous contact to control for tests (n = 50).

The sample size was calculated in the hypothesis of a conservative situation by comparing confirmed tuberculous participants (positive gold standard diagnostic test) and non -tuberculous (negative gold standard diagnostic test). The blood signature measured on venous blood samples showed a sensitivity of 93% in pregnant women. If the acceptable sensitivity for the new testing method is estimated at 96% and the prevalence of pulmonary TB in pregnant women in peripheral health centers is 12% and a precision of ± 7 is desired %and an α risk of 5%, a potency of 80%, the required sample size is 1167 pregnant women of which 140 are bacteriologically confirmed as active TB and 1027 controls. Considering an enrollment or rejection rate of 20%, the total needed sample would be 1,400 pregnant women in the CDT functions in the regions of Madagascar.

1. Data collection:

   Clinical data as well as biological samples (blood and sputum samples) are collected at the inclusion, the samples are analyzed at the Pasteur Institute of Madagascar.

   The data collection is done on paper based questionnaire where the data of each patient is recorded. The results of biological tests, paraclinical investigations as well as their results are also be recorded for each participant with the help of this questionnaire.
2. Data entry:

   The data are collected and transferred to a single database (REDCap). The REDCap system is compliant with the FDA standard CRF-21 part 11 as a reliable tool that allows to improve data quality and guarantee traceability. The data is stored on an IPM's secure server.
3. Data management and quality control:

   Data management is carried out by the IPM's Epidemiology and Clinical Research Unit (EPI-RC) data management team which closely collaborate with the study coordinators.

   Access to this database is restricted and secure. The list of persons with access rights appears in the data management manual. The data manager of the study is responsible for the security and quality of the data. A list of errors and inconsistencies detected in the database are regularly sent to the field team to make corrections. This regular monitoring will allow to improve the quality of the database. The request for partial or total extraction of the database must be the subject of a manuscript request and must have the consent of the epidemiological coordinator and scientific managers of the project.
4. Statistical analyzes:

   The entire study data is grouped into a single database and cleaned prior to any statistical processing of the data. All statistical analyzes will be performed on the GraphPad PRism and R software (http://www.R-project.org/) by designated competent persons for each data category studied.
5. Management of Potential Unnecessary Events:

   All undesirable events, observed during the study will be recorded in an observation register, which is either their severity and the link with the study procedures.

   Events will be coded using the 10th International Classification of Diseases (CIM-10) http://apps.who.int/classifications/icd10/browse).
6. Quality assurance:

Project investigators ensure the internal monitoring of the project at the study sites and are directly responsible for the collection, storage and transportation of the samples. Experienced laboratory technologists are in charge of manipulating and preparing samples for qPCR and DBS techniques at IPM.

Investigators and coordinators ensure that:

* the protocol is followed
* the recruitment of participants is done according to the planned schedule;
* Biological samples are labeled appropriately and consistently;
* the data is coherent and collected, recorded and secured as indicated in the data management plan of the study

The Coordinator and supervisors, recruited by the IPM, plan to visit the study sites regularly and is authorized to inspect the study documents so that patient confidentiality is maintained, in accordance with local regulations. The investigator cooperates with the coordinator so that any problems are identified during these control visits or resolved.

IPM has specific quality controls and assurance procedures developed and maintained in its laboratories and research units.

ELIGIBILITY:
Inclusion Criteria:

1. Group cases:

   * pregnant women aged over 15 adressed to TB diagnostic and treatment centers for a bacteriological diagnosis of pulmonary TB
   * Or with one or more symptoms of presumptive TB: cough, fatigue, weight loss, fever, chills, night sweats, shortness of breath, loss of appetite
   * agreed to participate in the study with full knowledge of the facts and signed an informed consent
2. Group control:

   * pregnant women over 15 years referred to a prenatal health center,
   * without known or clinically observed pathology associated with pregnancy
   * agreed to participate in the study with full knowledge of the facts and signed an informed consent

Exclusion Criteria:

1. Group cases :

   * Patients undergoing TB treatment for more than 2 weeks
   * Treatments with immunosuppressive drugs (≥ 14 consecutive days);
   * Progressive disease which does not allow venous blood sampling and venous capillary sampling;
   * All other clinical manifestations deemed incompatible for the study
2. Group Control :

   * No clinical signs of TB, no history of previous TB
   * No other known or clinically observed pathologies

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: All pregnant women addressed to 101 TB diagnostic and treatment centers of Madagascar
Sampling Method: Non-Probability Sample
Enrollment: 1424 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
diagnostic feature of test 3 G q-PCR capillary blood compared to gold stantard test | at inclusion
  The diagnostic performance are estimated by the sensitivity and specificity of the 3G q-PCR test with capillary blood compared to the sputum test as gold standard
diagnostic feature of test 3 G q-PCR capillary blood compared to 3 G q-PCR veinous blood | at inclusion
  The diagnostic performance are estimated by the sensitivity and specificity of the 3G q-PCR test with capillary blood compared to the 3 G q-PCR veinous blood as a reference test

CONTACTS AND LOCATIONS:
Overall Officials: Niaina RAKOTOSAMIMANANA, PhD, Principal Investigator — Institut Pasteur Madagascar
Locations (12):
- Madagascar (12):
  - CHRR Ambositra, CDT Ivato, Ambositra, Amoron'i Mania Region
  - CSBII Ivato, AMIT Behoririka, OSTIE Behoririka, CSB II Tanjombato, CSB II Analamahitsy, Antananarivo, Analamanga Region
  - CSB II Isotry Central, Dispensaire SALFA 67 ha, Centre Hospitalier d'Ambohidroa, Antananarivo, Analamanga Region
  - CSBII Ambohimanarina, CSB II Anosipatrana, CSB II Ambohipo, CHRD Itaosy, Antananarivo, Analamanga Region
  - Dispensaire SALFA Ambohibao, Centre Hospitalier de Soavinandriana, Dispensaire ECAR Anatihazo Isotry,, Antananarivo, Analamanga Region
  - Service de Pneumo-phtisio CHU Befelatanana, CHU de Soins et Santé Publique Analakely (CHUSSPA), Antananarivo, Analamanga Region
  - CHU Fenoarivo, Fenoarivo, Analamanga Region
  - DAT Toliara, SALFA Betela Toliara, Service Pneumo du CHU Toliara, Clinique Saint Luc, Toliara, Atsimo-Andrefana Region
  - DAT Toamasina, CHU PPH Toamasina, SALFA Toamasina, CSBII Foulpointe, Toamasina, Atsinanana Region
  - DAT Mahabibo, SALFA Antanimalandy, Service de Pneumologie CHU Androva, Mahajanga, Boeny Region
  - Service Pneumo du CHU Fianarantsoa, SALFA Ivory Atsimo, CHRD1 Ambohimahasoa, CHRD1 Ambalavao, Fianarantsoa, Upper Matsiatra
  - CHRR Antsirabe, SALFA Andranomadio, CSB II Mandoto, CSB II Ambohibary , CSB II Ambohibary, Antsirabe, Vakinankaratra Region

IPD SHARING:
Plan to Share IPD: Undecided
At the time of submission to the ethics committee, it will be decided to make a plan a share IPD

REFERENCES:
- [Background] Sweeney TE, Braviak L, Tato CM, Khatri P. Genome-wide expression for diagnosis of pulmonary tuberculosis: a multicohort analysis. Lancet Respir Med. 2016 Mar;4(3):213-24. doi: 10.1016/S2213-2600(16)00048-5. Epub 2016 Feb 20. PMID 26907218
- [Background] Sharma A, Jaiswal S, Shukla M, Lal J. Dried blood spots: concepts, present status, and future perspectives in bioanalysis. Drug Test Anal. 2014 May;6(5):399-414. doi: 10.1002/dta.1646. Epub 2014 Apr 1. PMID 24692095
- [Background] McAllister G, Shepherd S, Templeton K, Aitken C, Gunson R. Long term stability of HBsAg, anti-HBc and anti-HCV in dried blood spot samples and eluates. J Clin Virol. 2015 Oct;71:10-7. doi: 10.1016/j.jcv.2015.07.303. Epub 2015 Jul 29. PMID 26370308
- [Result] Rakotosamimanana N, Raharimanga V, Andriamandimby SF, Soares JL, Doherty TM, Ratsitorahina M, Ramarokoto H, Zumla A, Huggett J, Rook G, Richard V, Gicquel B, Rasolofo-Razanamparany V; VACSEL/VACSIS Study Group. Variation in gamma interferon responses to different infecting strains of Mycobacterium tuberculosis in acid-fast bacillus smear-positive patients and household contacts in Antananarivo, Madagascar. Clin Vaccine Immunol. 2010 Jul;17(7):1094-103. doi: 10.1128/CVI.00049-10. Epub 2010 May 12. PMID 20463103
- [Result] Ostler MW, Porter JH, Buxton OM. Dried blood spot collection of health biomarkers to maximize participation in population studies. J Vis Exp. 2014 Jan 28;(83):e50973. doi: 10.3791/50973. PMID 24513728
- [Result] Gruner N, Stambouli O, Ross RS. Dried blood spots--preparing and processing for use in immunoassays and in molecular techniques. J Vis Exp. 2015 Mar 13;(97):52619. doi: 10.3791/52619. PMID 25867233